CLINICAL TRIAL: NCT02584933
Title: An Open-label, Multi-center, Phase IV Roll-over Study in Patients With ALK Positive Malignancies Who Have Completed a Novartis-sponsored Ceritinib (LDK378) Study and Are Judged by the Investigator to Benefit From Continued Treatment With Ceritinib
Brief Title: Roll-over Study to Allow Access to Certinib (LDK378) for Patients Who Are on Ceritinib Treatment in a Novartis-sponsored Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2X01B; 2024-511040-58-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT01947608 (No longer available)
Record Dates: First submitted 2015-10-06; First posted 2015-10-23 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: ALK Positive Malignancies
Keywords: ALK; Malignancies
MeSH Terms: conditions — Neoplasms | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ceritinib (Experimental): The starting dose of study treatment for patients in this protocol should be the same as the dose provided in the parent ceritinib study at the time of the rollover.
  Interventions: Drug: ceritinib

INTERVENTIONS:
Drug: ceritinib — hard gelatin capsule or hard tablet for oral use up to 750 mg

SUMMARY:
The rollover study will provide ceritinib to patients who are currently receiving treatment with ceritinib within a Novartis-sponsored study and in the opinion of the investigator, would benefit from continued treatment with ceritinib.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently receiving treatment with ceritinib within a Novartis-sponsored study which has fulfilled the requirements for the primary objective and, in the opinion of the Investigator, would benefit from continued treatment.
* Patient has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements.
* Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures.
* Written informed consent obtained prior to enrolling in the roll-over study and receiving study medication. If consent cannot be expressed in writing, it must be formally documented and witnessed via an independent trusted witness.

Exclusion Criteria:

* Patient has been permanently and prematurely discontinued from ceritinib study treatment in the parent study due to any reason.
* Patient currently has unresolved toxicities for which ceritinib dosing has been interrupted in the parent study.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months afer stopping ceritinib treatment.
* Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after stopping ceritinib and should not father a child for at least 3 months after the last dose of treatment.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Until no patients are left on study up to 5 years
  To collect safety data: adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- United States (5):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Loma Linda University, Loma Linda, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Maryland Oncology Hematology P A, Rockville, Maryland
  - Essex Oncology of North Jersey PA, Belleville, New Jersey
- Australia (2):
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Auckland
- Novartis Investigative Site, Leuven, Belgium
- Brazil (4):
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sofia, Bulgaria
- China (4):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
- Novartis Investigative Site, Montería, Colombia
- Novartis Investigative Site, Brno, Czechia
- France (4):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Villejuif
- Germany (5):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (12):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Koto Ku, Tokyo
- Novartis Investigative Site, Beirut, Lebanon
- Malaysia (2):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kuching, Sarawak
- Novartis Investigative Site, Gdansk, Poland
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District